CLINICAL TRIAL: NCT05954260
Title: Cuantificación de la Disfunción Inmunitaria Inducida Por la Enfermedad Crítica Mediante el Estudio de un Panel de Genes y Moléculas Implicadas en la Sinapsis Inmunológica y su Utilidad Pronóstica
Brief Title: Immune Dysfunction in Critical Illness: Utility of a Panel of Genes and Molecules Involved in the Immunological Synapse
Acronym: EFIMERO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: David Pérez Torres (Other)
Collaborators: Hospital del Rio Hortega (Other); Sanidad de Castilla y León (Other); Instituto de Investigación Biomédica de Salamanca (Other); Fundación Española del Enfermo Crítico (FEEC) (Unknown); Sociedad Española de Medicina Intensiva, Crítica y Unidades Coronarias (SEMICYUC) (Unknown)
Responsible Party: Sponsor-Investigator, David Pérez Torres, Principal Investigator, University of Valladolid
Organization: University of Valladolid (Other)
Other Study IDs: EFIMERO; FEEC 2022/001 (Other Grant/Funding Number: SEMICYUC); GRS 2618/A/22 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y León (SACYL))
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Critical Illness
Keywords: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect blood samples from the patients included in the study on ICU days 1, 3 and 5. We will measure gene expression (mRNA) and plasma levels of various elements involved in the immunological synapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sampling — We will collect blood samples from the patients included in the study on ICU days 1, 3 and 5. We will measure gene expression (mRNA) and plasma levels of various elements involved in the immunological synapse.

SUMMARY:
Critical illnesses represent a significant physiological assault that triggers changes in the patient's immune system, resulting in an immunopotentiating response (systemic inflammatory response syndrome, SIRS) and an immunosuppressive response (compensatory anti-inflammatory response syndrome, CARS). The balance between SIRS and CARS is essential for the patient to return to a state of immune homeostasis and accelerate the healing process. However, when CARS is disproportionately intense, it leads to a state of immunoparalysis, which predisposes the patient to vulnerability to opportunistic infections, associated with a peak in late mortality. The majority of patients admitted to the ICU are considered immunocompetent. However, the investigators suspect that a significant proportion of them exhibit predominance of CARS and a state of functional immunosuppression. There is currently no diagnostic test to determine whether a patient is functionally immunocompetent at a specific point in time.

The goal of this observational study is to learn about the immune system dysfunction occurring in critical illness. The main questions it aims to answer are:

* What is the prevalence of immune system dysfunction in critical illness?
* Does immune system dysfunction affect multiple organ failure trajectory and mortality in critical illness?
* Is immune system dysfunction related to an increased risk of opportunistic hospital-acquired infections in critical illness?
* Is immune system dysfunction related to age, fragility, nutritional status or previous comorbidities in critical illness?

To answer these questions, the investigators will prospectively study a population of critically ill patients, defined by the presence of organ failure. The investigators will analyse a panel of genes and molecules involved in immunological synapse, using peripheral blood samples at different moments of the evolution of critical illness. Based on the analysis, the investigators will classify the patients' functional immune status and correlate it with the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Failure of one or more organs, assessed by a Sequential Organ Failure Assessment Score (SOFA) ≥4 within the first 24 hours of admission to the Intensive Care Unit (ICU). At least one of the physiological systems involved must be in the category of organ failure and, therefore, score ≥3.
* Informed consent to participate in the study.
* Age equal to or greater than 18 years.

Exclusion Criteria:

* Pharmacological immunosuppression within the 3 months prior to the current admission date, including treatment with corticosteroids, immunosuppressive drugs (conventional or biological), or chemotherapy.
* Immunodeficiency.
* Age under 18 years.
* Absence of consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any critical illness present in the ICU of the participating hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse.
Mortality (28-day) | 28 days
  Number of non-surviving patients in the groups with and without an early functional immunosuppression signature.
Hospital-Acquired Infection (28-day) | 28 days
  Number of patients developing hospital-acquired infections in the groups with and without an early functional immunosuppression signature.
Organ Failure Resolution (28-day) | 28 days
  Number of patients with organ failure resolution in the groups with and without an early functional immunosuppression signature.

SECONDARY OUTCOMES:
Mortality (90-day) | 90 days
  Number of non-surviving patients in the groups with and without an early functional immunosuppression signature.
Hospital-Acquired Infection (90-day) | 90 days
  Number of patients developing hospital-acquired infections in the groups with and without an early functional immunosuppression signature.
Duration of hospitalization in the ICU | 90 days
  Length of stay in the ICU in the groups with and without an early functional immunosuppression signature.
Proportion of patients requiring organ support | 90 days
  Number of patients who require organ support (mechanical ventilation, vasopressors, renal replacement therapy, extracorporeal membrane oxygenation,...) in the groups with and without an early functional immunosuppression signature.
Proportion of patients with early cardiac dysfunction | 5 days
  Number of patients who develop early cardiac dysfunction, as assessed by echocardiography, in the groups with and without an early functional immunosuppression signature.
Proportion of patients with Herpesviridae reactivation | 90 days
  Number of patients who develop Herpesviridae reactivation during ICU admission, in the groups with and without an early functional immunosuppression signature.
Proportion of patients with ICU-related complications | 90 days
  Number of patients who develop ICU-related complications during ICU admission, including ICU-acquired weakness, delirium, thrombosis or bleeding, in the groups with and without an early functional immunosuppression signature.
Proportion of patients with post-intensive care syndrome | 90 days
  Number of patients who develop post-intensive care syndrome, in the groups with and without an early functional immunosuppression signature.

OTHER OUTCOMES:
Sex-related differences in the proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse, grouped by sex category.
Age-related differences in the proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse, grouped by predefined age categories.
Nutritional status-related differences in the proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse, grouped by nutritional status on ICU admission.
Frailty status-related differences in the proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse, grouped by frailty status on ICU admission.
Comorbid status-related differences in the proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse, grouped by previous comorbidities.
Diagnosis-related differences in the proportion of patients with a functional immunosuppression signature | 5 days
  Number of patients with organ failure exhibiting an early transcriptomic signature denoting depression of the immunological synapse, grouped by diagnostic category on ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: David Pérez-Torres, MD, Principal Investigator — Hospital Universitario Río Hortega, Universidad de Valladolid
Locations (1):
- Hospital Universitario Río Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided